CLINICAL TRIAL: NCT04466319
Title: The Effect of Rocking Chair Movement on the Start of Bowel Functions in Patients With Gastrointestinal System Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Yasemin Şara, research assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 80558721-050.99-E.25047
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Ileus
Keywords: Ileus; Gastrointestinal Diseases; Gastrointestinal Motility; Postoperative Complications; Nurses
MeSH Terms: conditions — Ileus; Gastrointestinal Diseases; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study in patients with open gastrointestinal tract surgery to evaluate the effect of rocking chair movement to be given in addition to standard care at the start of postoperative bowel functions (post-operative first gas, initial defecation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): The individuals in the intervention group in the rocking chair three times a day, 20 minutes, a total of 60 minutes after the first day after surgery.They did this intervention until they first defecation .
  Interventions: Other: Rocking Chair
- Control arm (No Intervention): The individuals in the control group sat in a standard chair in the same time as the intervention group in the non-rocking chair.

INTERVENTIONS:
Other: Rocking Chair — Patients in the experimental group were sat rocking chair three times a day in a rocking wooden chair in addition to their postoperative routine care by their nurses. After providing the rocking chair to the patients' room, the researcher gave the data collection form to be filled by the patient himself. It was the researcher's supervision that the patient sat in the rocking chair for the first time. The rocking chair movement continued to intervene until the patient released gas. After emitting gas, he continued to swing in the rocking chair until he made his first stools. The patient was visited every day until he was discharged. No special clothing or materials were required for the patients to sit in the rocking chair.
  Arms: intervention arm

SUMMARY:
The Effect of Rocking Chair Movement on the Start of Bowel Functions in Patients With Gastrointestinal System Surgery

The research will be carried out as a randomized controlled experimental study in patients with open gastrointestinal tract surgery in order to evaluate the effect of rocking chair movement to be given in addition to standard care in the initiation of postoperative bowel functions (post-operative first time gas, first time defecation).Ethics committee and institution permissions and written consents of individuals were obtained prior to the study.The universe of the study was composed of patients with open gastrointestinal surgery lying in the general surgery service of a hospital in Eskisehir. With the error margin of 0.05, 90% test power, 30 people in intervention and control groups, 60 patients in total will be included in the research.Appointment of patients to intervention and control groups was done by stratification and block randomization method according to gastric and intestinal surgery.The draw method was used to assign stratified patients to blind technique intervention and control groups in order to avoid side-holding, and an equal number (blocking) patients were assigned to each group. The individuals in the intervention group in the rocking chair three times a day, 20 minutes, a total of 60 minutes after the first day after surgery. The individuals in the control group will sit in a standard chair in the same time as the intervention group in the non-rocking chair. The data will be collected using the "Descriptive characteristics determination form", "Intervention Group Intestinal Functions Evaluation Form" and "Control Group Intestinal Functions Evaluation Form".

DETAILED DESCRIPTION:
Inclusion Criteria

* Accepting to participate in the research
* Being 18 or over
* Having gastrointestinal surgery
* No communication problems
* No symptoms or disease (dizziness, Vertigo, Meniere.) That rocking chair movement will adversely affect the patient
* With or without a stoma in the postoperative period;
* Patients with ASA (American Society of Anesthesiology) classification I or II

Exclusion Criteria

* Not agreeing to participate in the research
* Being 18 or under
* Being a communication problem
* The symptoms or disease (dizziness, Vertigo, Meniere.) That the rocking chair movement will adversely affect the patient.
* Having a history of ileus after surgery
* Any complication after surgery
* With inflammatory and irritable bowel disease
* Using drugs that will affect intestinal motility before or after surgery.
* Surgical intervention is laparoscopic
* ASA classification is III, IV or V

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the research
* Being 18 or over
* Having gastrointestinal surgery
* No communication problems
* No symptoms or disease (dizziness, Vertigo, Meniere.) That rocking chair movement will adversely affect the patient With or without a stoma in the postoperative period;
* Patients with American Society of Anesthesiology (ASA) classification I or II

Exclusion Criteria:

* Not agreeing to participate in the research
* being 18 or under
* Being a communication problem
* The symptoms or disease (dizziness, Vertigo, Meniere.) That the rocking chair movement will adversely affect the patient.
* Having a history of ileus after surgery
* Any complication after surgery
* With inflammatory and irritable bowel disease
* Using drugs that will affect intestinal motility before or after surgery.
* Surgical intervention is laparoscopic
* ASA classification is III, IV or V

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
time to report of first flatus | Defined as the first time hear the bowel sound after surgery1-5 days
  Defined as the first time flatus happens
time to report of first defecation | End of surgery to the first defecation 1-7 days
  Defined as the first time defecation happens.

SECONDARY OUTCOMES:
length of postoperative hospitalization | End of surgery to hospital discharge 5-7 days
  Defined as the length hospitalization after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nedime Köşgeroğlu, Prof, Study Director — T.C. İstanbul Rumeli University
Locations (1):
- Dean of the Faculty of Medicine Ground Floor Meşelik Campus, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No